CLINICAL TRIAL: NCT03714568
Title: Pharmacokinetic and Tolerance Study in Healthy Participants: a Single-centre, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Pharmacokinetic and Tolerance Study of TQ-A3326 in Healthy Participants.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ZDTQ-A3326-1
Record Dates: First submitted 2018-05-28; First posted 2018-10-22 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-07

CONDITIONS: Pharmacokinetic
MeSH Terms: interventions — TQ-A3326

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ-A3326 (Experimental): TQ-A3326 (15mg-180mg: p.o. single dose; 60mg: p.o. multi-doses）
  Interventions: Drug: TQ-A3326
- placebo (Experimental): Placebo(15-180mg: p.o. single dose; 60mg: p.o. multi-doses)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: TQ-A3326 — TQ-A3326 (15mg-180mg: p.o. single dose; 60mg: p.o. multi-doses）
  Arms: TQ-A3326
Drug: placebo — Placebo(15-180mg: p.o. single dose; 60mg: p.o. multi-doses)
  Arms: placebo

SUMMARY:
To study the single dose and multi-doses pharmacokinetic characteristics and tolerance of TQ-A3326 in the human body；To study the transformation of TQ-A3326；To study the effect of the food on the pharmacokinetic characteristics of TQ-A3326.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, age 18 to 60 years, inclusive.
* The body weight of male is not less than 50kg, and female is not less than 45kg. All participants' body mass index (BMI) is between 19~26.
* Adequate blood cell counts, kidney function and liver function.
* Healthy participants should participate in the study voluntarily and sign informed consent.

Exclusion Criteria:

* Subjects with known allergy to the similar products tested.
* Subject is on a special diet (for example subject is vegetarian).
* Medical demographics with evidence of clinically significant deviation from normal medical condition.
* Female subjects who were pregnant or nursing.
* Results of laboratory tests which are clinically significant.
* Acute infection within one week preceding first study drug administration.
* History of drug or alcohol abuse.
* Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
* Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
* ale subjects (or their partner) or female subjects have the unprotective sex behavior or have a planned pregnancy during the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Serious Adverse Events (SAEs). | Day 1 up to Day 7 for non-SAEs .
  SAEs were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Number of Participants With Clinically Significant Change From Baseline in Vital Sign Measurements. | Day 1 up to Day 7 or Discharge.
  Participants were assessed by investigator for any clinically significant changes in vital parameters like body temperature, respiratory rate, blood pressure, heart rate and weight. The assessment was performed by a calibrated sphygmomanometer and thermometer for blood pressure and temperature, respectively. Blood pressure and heart rate were measured after at least 5 minutes quiet seating of the subject. Weight was measured at the discharge. The criteria for clinically significant change was as per the investigators discretion.
Number of Participants With Marked Abnormalities in Laboratory Findings. | Day 1 up to Day 7.
  Laboratory marked abnormalities were defined as Hematocrit (low) as <0.85*pre-treatment value, Leukocytes (low) as <0.9*lower limit of normal, Aspartate Aminotransferase (high) as >1.25*upper limit of normal, Creatinine (high) as >1.33*pre-treatment value, Bicarbonate (high) as >1.2*upper limit of normal, Total Protein (high) as >1.1*upper limit of normal, Creatinine Kinase (high) as >1.5*upper limit of normal, Blood in Urine (high) as ≥ 2*upper limit of normal. Participants were fasted for at least 10 hours prior to the collection of blood specimens for clinical laboratory tests.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax). | Pre-dose, 0.25hour, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour, 72hour, 96hour, 120hour post-dosing on Day 1
  Maximum observed plasma concentration following drug administration from the raw plasma concentration-time data. The plasma samples were analyzed for TQ-A3326 using a validated liquid chromatography-tandem mass spectrometric assay.
  2）Grade 4 hematology toxicity
Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC[0-T]). | Pre-dose, 0.25hour, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour, 72hour, 96hour, 120hour post-dosing on Day 1.
  Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration. It was calculated as the sum of linear trapezoids using non-compartmental analysis. The plasma samples were analyzed for TQ-A3326 using a validated liquid chromatography-tandem mass spectrometric assay.
Area Under the Plasma Concentration-time Curve From Time Zero (AUC[INF]) Extrapolated to Infinite Time. | Pre-dose, 0.25hour, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour, 72hour, 96hour, 120hour post-dosing on Day 1.
  Area under the plasma concentration-time curve from time zero extrapolated to infinite time was estimated as sum of AUC(0-T) and the extrapolated area, computed by the quotient of the last observable concentration and λ, where λ was the slopes of the terminal phases of the plasma concentration-time profiles. The plasma samples were analyzed for TQ-A3326 using a validated liquid chromatography-tandem mass spectrometric assay.
Time to Reach Maximum Plasma Concentration (Tmax). | Pre-dose, 0.25hour, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour, 72hour, 96hour, 120hour post-dosing on Day 1.
  Tmax was defined as the time required to reach maximum observed plasma concentration. The plasma samples were analyzed for TQ-A3326 using a validated liquid chromatography-tandem mass spectrometric assay.
Plasma Half-life (T-half) | Pre-dose, 0.25hour, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour, 72hour, 96hour, 120hour post-dosing on Day 1.
  Plasma half-life was defined as the time required for one half of the total amount of administered drug eliminated from the body. The plasma samples were analyzed for TQ-A3326 using a validated liquid chromatography-tandem mass spectrometric assay.
Apparent Total Body Clearance (CLT/F) | Pre-dose, 0.25hour, 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 6hour, 8hour, 12hour, 24hour, 48hour, 72hour, 96hour, 120hour post-dosing on Day 1.
  Apparent total body clearance (CLT/F) was calculated as Dose/AUC(INF), where CLT was the clearance of the drug and F was the absolute oral bioavailability. The plasma samples were analyzed for TQ-A3326 using a validated liquid chromatography-tandem mass spectrometric assay.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided